CLINICAL TRIAL: NCT02798107
Title: Safety of Potential Paediatric Patients Treated With Idarucizumab: a Non-internventional Chart Review Study
Brief Title: Observational Study to Evaluate Safety of Idarucizumab in Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1321.11
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients treated with idarucizumab
  Interventions: Drug: idarucizumab

INTERVENTIONS:
Drug: idarucizumab — drug

SUMMARY:
Idarucizumab is a humanized monoclonal antibody fragment (Fab) that binds to dabigatran with very high affinity. Idarucizumab potently and specifically binds to dabigatran and its metabolites and neutralises its anticoagulant effect. A clinical development program is ongoing to support marketing authorisation submissions for idarucizumab indicated in patients treated with dabigatran who require emergency surgery/urgent procedures or who have a life-threatening or uncontrolledbleeding when rapid reversal of the anticoagulant effects of dabigatran is required.

DETAILED DESCRIPTION:
Purpose:

Study Design:

ELIGIBILITY:
Inclusion criteria:

* Male or female, <18 years of age
* Were administered idarucizumab at sites and usage identified by various methods (eg.through the Idarucizumab drug administration surveillance program, spontaneous reporting)

Exclusion criteria:

Participation in a dabigatran or idarucizumab clinical trial

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any pediatric patient who has received a commercial supply of idarucizumab following market approval in their country
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2019-05-23 (Estimated); Study Completion 2019-05-24 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes until hospital discharge * Incidence of thromboembolic events (ie. obstruction of a blood vessel by the formation of a thrombus - e.g. ischemic stroke, MI, DVT, PE) after administration | Up to 33 months
Safety outcomes until hospital discharge * Incidence of hypersensitivity/anaphylactic reactions | Up to 33 months
Safety outcomes until hospital discharge * Incidence of AE, SAE, ADR, SADR reporting | Up to 33 months
Safety outcomes until hospital discharge * Cause of death and in-hospital mortality rate | Up to 33 months

SECONDARY OUTCOMES:
Comparison of patient characteristics of paediatric patients with & without outcome events * Incidence of thromboembolic events (ie. obstruction of a blood vessel by the formation of a thrombus - e.g. ischemic stroke, MI, DVT, PE) after administration | Up to 33 months
Comparison of patient characteristics of paediatric patients with & without outcome events * Incidence of hypersensitivity/anaphylactic reactions | Up to 33 months
Comparison of patient characteristics of paediatric patients with & without outcome events * Incidence of AE, SAE, ADR, SADR reporting | Up to 33 months
Comparison of patient characteristics of paediatric patients with & without outcome events * Cause of death and in-hospital mortality rate | Up to 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing